CLINICAL TRIAL: NCT07300566
Title: FOcal Versus Whole Gland High Dose-Rate Brachytherapy (HDR-BT) Boost With ExternAl Beam Radiotherapy in LocalizeD Prostate Cancer: A Phase 2 Randomized Trial [FORWARD]
Brief Title: Focal Versus Whole Gland High Dose-Rate Brachytherapy (HDR-BT) Boost to External Beam Radiotherapy in Localized Prostate Cancer: A Phase 2 Randomized Trial
Acronym: FORWARD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joelle Helou (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Joelle Helou, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORWARD - ReDA 16623
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Focal high dose rate brachytherapy; Whole gland high dose rate brachytherapy; External beam radiotherapy; Intermediate risk prostate cancer; High risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Gland High Dose Rate Brachytherapy Boost Arm (Active Comparator)
  Interventions: Radiation: Standard Arm: Whole Gland High Dose Rate Brachytherapy Boost
- Focal High Dose Rate Brachytherapy Boost Arm (Experimental)
  Interventions: Radiation: Experimental Arm: Focal High Dose Rate Brachytherapy Boost

INTERVENTIONS:
Radiation: Standard Arm: Whole Gland High Dose Rate Brachytherapy Boost — Whole gland high dose rate brachytherapy (15 Gray/1 fraction) plus stereotactic ablative radiotherapy to the prostate +/- pelvis (25 Gray/5 fractions). Androgen deprivation therapy 6 to 24 months (physician discretion).
  Arms: Whole Gland High Dose Rate Brachytherapy Boost Arm
Radiation: Experimental Arm: Focal High Dose Rate Brachytherapy Boost — Focal high dose rate brachytherapy boost to the dominant intraprostatic lesion (15 Gray/1 fraction) plus stereotactic ablative radiotherapy to the prostate (30 Gray/5 fractions) +/- the pelvis (25 Gray/5 fractions). Androgen deprivation therapy 6 to 24 months (physician discretion).
  Arms: Focal High Dose Rate Brachytherapy Boost Arm

SUMMARY:
This project aims to compare the changes in the urinary quality of life (QoL) following focal high dose-rate brachytherapy (HDR-BT) boost to stereotactic ablative radiotherapy (SABR), compared to standard whole gland HDR-BT boost, in the treatment of men diagnosed with intermediate- and high-risk prostate cancer, with have an identifiable DIL on mpMRI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* Eastern Co-Operative Oncology Group (ECOG) 0-2
* Intermediate and high-risk disease with localized unfavorable features:

  * defined as clinical stage tumor cT1 or cT2a, International Society of Urological Pathology (ISUP) grade group 2-4 in less than or equal to 50% of the cores, unilateral extracapsular extension (ECE), prostate specific antigen (PSA) less than or equal to 20 ng/mL
  * corresponding to an Identified dominant intraprostatic lesion (DIL) on multiparametric magnetic resonance imaging (mpMRI) Prostate Imaging Reporting and Data System score (PI-RADs 3-5)
* Prostate volume less than or equal to 60 cc is recommended. Transrectal ultrasound (TRUS) and magnetic resonance imaging (MRI) are accepted to assess prostate volume. Patients with a prostate volume between 60 and 80 cc can be included if the International Prostate Symptom Score (IPSS) is less than 15 and brachytherapy is deemed feasible by the treating physician.

Exclusion Criteria:

* Contraindications to mpMRI
* Documented nodal or distant metastases
* Previous pelvic radiotherapy
* Recent transurethral resection of prostate (less than or equal to 6 months), previous prostatectomy or high-intensity focused ultrasound (HIFU)
* Poor baseline urinary function: International Prostate Symptom Score (IPSS) greater than 19
* Connective tissue disease or inflammatory bowel disease
* Patients deemed unsuitable for general anaesthetic by the Anaesthesia Department
* Patient is unable to lie flat long enough for the Radiation Therapy (RT) Simulation and Treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Urinary Quality of Life at 24 Months Measured by the Expanded Prostate Index Composite (EPIC-26) Questionnaire | From enrollment to 24 months post radiation therapy
  To compare the impact on urinary quality of life (QoL) between focal high dose-rate brachytherapy (HDR-BT) boost and standard whole gland HDR-BT boost to stereotactic ablative radiotherapy (SABR) as reported by the participant on the Expanded Prostate Index Composite (EPIC-26) questionnaire.

SECONDARY OUTCOMES:
Acute Changes in Urinary, Bowel, and Sexual Quality of Life | Less than or equal to 6 months post radiation therapy
Long Term Changes in Bowel and Sexual Quality of Life Measured by Expanded Prostate Index Composite (EPIC-26) Questionnaire | From enrollment to 24 months post radiation therapy
  Changes in bowel and sexual health as reported by the participant on the Expanded Prostate Index Composite (EPIC-26) questionnaire.
Acute and Chronic Physician-Reported Toxicity Using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | From enrollment to 24 months post radiation therapy
  Severity and grade of side effects of treatment as reported by the physician using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Prostate Specific Antigen (PSA) at 4 years | 4 years post radiation therapy
  Blood test measuring the amount of PSA protein made by the prostate.
Biochemical Control Measure by Prostate Specific Antigen (PSA) Levels | Enrollment to 5 years post radiation therapy
Participant reported Symptoms Measured by the Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | From enrollment to 24 months post radiation therapy
  Frequency and severity of side effects of treatment as reported by the participant on the Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Joelle Helou, MD, Principal Investigator — London Health Sciences Centre Research Institute, London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, Verspeeten Family Cancer Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No